CLINICAL TRIAL: NCT00059345
Title: The Impact of Patient-Provider Interaction on Response to Acupuncture
Brief Title: Interaction Between Patient and Healthcare Provider: Response to Acupuncture in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR049999 (NIH); R01AR049999 (NIH); NIAMS-087 (Other: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)); 2006-0605 (Other: UT MDACC Study ID)
Record Dates: First submitted 2003-04-23; First posted 2003-04-24 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthritis
Keywords: Acupuncture; Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis | interventions — Acupuncture Therapy; Electroacupuncture; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Acupuncture (Experimental): Participants will receive acupuncture
  Interventions: Procedure: Acupuncture
- Arm 2: Shallow needling (Placebo Comparator): Participants will receive shallow needling on non-mederian points
  Interventions: Procedure: Placebo acupuncture
- Arm 3: No Acupuncture or Placebo Treatment (Other): Participants will receive usual care, no acupuncture or placebo acupuncture treatment.
  Interventions: Other: Usual Care

INTERVENTIONS:
Procedure: Acupuncture — Electroacupuncture treatments provided two times per week for 6 weeks
  Other Names: Electroacupuncture; TENS
  Arms: Arm 1: Acupuncture
Procedure: Placebo acupuncture — Placebo acupuncture treatments provided 2 times per week for 6 weeks
  Other Names: Sham acupuncture
  Arms: Arm 2: Shallow needling
Other: Usual Care — Usual care for knee osteoarthritis
  Arms: Arm 3: No Acupuncture or Placebo Treatment

SUMMARY:
Interactions between patients and healthcare providers may have a significant impact on a patient's response to therapy. In this study, patients with osteoarthritis (OA) of the knee will receive either acupuncture or sham acupuncture. The acupuncturists will be trained to interact with the patients in specific ways. The study will evaluate those interactions.

DETAILED DESCRIPTION:
This study will examine placebo responses in the context of practitioner-patient interactions at the time of the encounter. Phase 1 of this study identified patient-related determinants of placebo response, such as beliefs and expectations toward treatment of knee OA with acupuncture. Phase 2 of the study evaluated an assessment tool to measure these determinants. Phase 3 of the study is a randomized controlled trial to evaluate whether placebo effects in patients with knee OA can be enhanced by the acupuncturists' communicative style, which can affect a patient's cognitive expectancies and beliefs.

Patients will initially be randomized to one of two groups, each with a different model for practitioner-patient interaction. Acupuncture practitioners will be trained to follow semi-structured communicative styles, including traditional approaches in Chinese medicine and techniques previously described in patient-doctor communications studies. Within each of these groups, patients will be further randomized to receive either acupuncture or sham acupuncture. Patients will have 6 weeks of biweekly treatment visits. Patients will be followed for 6 months. Visits will be weekly during the first 6 weeks of the study and monthly thereafter.

The study will also include a natural cohort group composed of patients on a study waiting list; these patients will be offered acupuncture 3 months after study entry.

ELIGIBILITY:
Inclusion Criteria:

* OA diagnosis according to the American College of Rheumatology criteria
* Pain in the knee of at least 3 or more on a 0 to 10 scale (0 none, 10 extreme pain) within 2 weeks prior to study entry
* Stable treatment with anti-inflammatory and analgesic medications during the month prior to study entry
* If receiving glucosamine, stable dosage for 2 months prior to study entry
* Adequate cognitive status as determined by the study officials
* Living in the community
* Ability to communicate in English without a translator
* Access to a telephone

Exclusion Criteria:

* Other diagnosed joint diseases, such as rheumatoid arthritis
* Previous treatment with acupuncture (for any condition)
* Intra-articular injections in the knee in the 2 months prior to study entry

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2002-09; Primary Completion 2006-07 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale | 3-month
Joint-Specific Multidimensional Assessment of Pain (J-MAP) to evaluate placebo effects on the different dimensions of pain | 3-month
Patient satisfaction with their knee condition (SKIP) | 3-month

SECONDARY OUTCOMES:
SF-12 | 3-month
Range of motion of each knee | 3-month
Timed walking test | 3-month
Locus of control | Baseline
Optimism | 3-month
Self-efficacy | baseline
Cognitive pain | 3-month
Anxiety | 3-month
Social support | 3-month
Patient reaction | 3-month
Physician trust | 3-month

CONTACTS AND LOCATIONS:
Overall Officials: Maria E. Suarez-Almazor, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Suarez-Almazor ME, Looney C, Liu Y, Cox V, Pietz K, Marcus DM, Street RL Jr. A randomized controlled trial of acupuncture for osteoarthritis of the knee: effects of patient-provider communication. Arthritis Care Res (Hoboken). 2010 Sep;62(9):1229-36. doi: 10.1002/acr.20225. PMID 20506122
- [Derived] Street RL Jr, Cox V, Kallen MA, Suarez-Almazor ME. Exploring communication pathways to better health: clinician communication of expectations for acupuncture effectiveness. Patient Educ Couns. 2012 Nov;89(2):245-51. doi: 10.1016/j.pec.2012.06.032. Epub 2012 Jul 31. PMID 22857778
- See also: University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org